CLINICAL TRIAL: NCT04049266
Title: A Phase 2b/3, Prospective, Randomized, Double-masked, Active Comparator-controlled, Multi-center Study to Investigate the Efficacy and Safety of Repeated Intravitreal Administration of KSI-301 in Subjects With Neovascular (Wet) Age-related Macular Degeneration.
Brief Title: A Study to Evaluate the Efficacy and Safety of KSI-301, an Anti-VEGF Antibody Biopolymer Conjugate, Versus Aflibercept in Patients With Neovascular (Wet) Age-Related Macular Degeneration.
Acronym: DAZZLE
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Primary Endpoint Not Met
Sponsor: Kodiak Sciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KSI-CL-102
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-06

CONDITIONS: Wet Macular Degeneration
Keywords: AMD; Wet AMD; choroidal neovascularization secondary to age-related macular degeneration; KSI-301; Aflibercept; Vascular endothelial growth factor; VEGF; Anti-VEGF; Antibody biopolymer conjugate; Macular Degeneration; Wet Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases; Vision Disorders; Vision, low; Kodiak
MeSH Terms: conditions — Wet Macular Degeneration; Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases; Vision Disorders; Vision, Low | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A masked evaluating investigator will be responsible for subject care except the injections and the safety assessment following the injections. An unmasked treating investigator will perform the injections and assess patient safety following the injections.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KSI-301 5 mg (Experimental): Drug: KSI-301 5 mg. KSI-301 5 mg will be administered by intravitreal injection into the study eye at 12, 16, and 20 weeks intervals as specified in the study protocol.
  Drug: Sham Procedure. The sham is a procedure that mimics an intravitreal injection. It involves pressing the blunt end of an empty syringe (without a needle) against the anesthetized eye. It will be administered to participants in both treatments arms at applicable visits to maintain masking.
  Interventions: Drug: KSI-301; Other: Sham Procedure
- Aflibercept 2 mg (Active Comparator): Drug: Aflibercept 2 mg. Aflibercept 2 mg will be administered by intravitreal injection into the study eye once every 4 weeks for 3 consecutive months, followed by once every 8 weeks.
  Drug: Sham Procedure. The sham is a procedure that mimics an intravitreal injection. It involves pressing the blunt end of an empty syringe (without a needle) against the anesthetized eye. It will be administered to participants in both treatments arms at applicable visits to maintain masking.
  Interventions: Drug: Aflibercept; Other: Sham Procedure

INTERVENTIONS:
Drug: KSI-301 — Intravitreal Injection
  Arms: KSI-301 5 mg
Drug: Aflibercept — Intravitreal Injection
  Other Names: Eylea
  Arms: Aflibercept 2 mg
Other: Sham Procedure — The sham is a procedure that mimics an intravitreal injection. It involves pressing the blunt end of an empty syringe (without a needle) against the anesthetized eye. It will be administered to participants in both treatments arms at applicable visits to maintain masking.

SUMMARY:
This study will evaluate the efficacy, safety, durability, and pharmacokinetics of KSI-301 administered at 12, 16 and 20 weeks intervals as specified in the protocol, compared with aflibercept once every 8 weeks (Q8W), in participants with treatment-naïve neovascular (wet) age-related macular degeneration (nAMD).

DETAILED DESCRIPTION:
This study is divided into a 3-week screening period, a 92-week treatment period, and a final 4-week follow-up period. At baseline patients will be randomized 1:1 into two treatment arms: KSI-301 5 mg and aflibercept 2 mg.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to participation in the study.
* Active, treatment-naïve choroidal neovascularization (CNV) secondary to AMD.
* BCVA ETDRS score between 80 and 25 letters (Snellen equivalent of 20/25 to 20/320), inclusive.
* Other protocol-specified inclusion criteria may apply

Exclusion Criteria:

* CNV secondary to other causes in the Study Eye.
* Any history of macular pathology unrelated to AMD but affecting vision or contributing to subretinal or intraretinal fluid.
* Any history or evidence of a concurrent intraocular condition in the Study Eye that, in the judgment of the Investigator, could require either medical or surgical intervention during the study to prevent or treat visual loss.
* Active ocular or periocular infection or inflammation.
* Prior administration of any approved or investigational treatment for neovascular AMD in the Study Eye.
* Uncontrolled glaucoma in the Study Eye.
* Women who are pregnant or lactating or intending to become pregnant during the study.
* Stroke or myocardial infarction in the 6-month period prior to Day 1.
* Uncontrolled blood pressure defined as a systolic value > 180 mmHg or diastolic value ≥100 mmHg while at rest.
* History of a medical condition that, in the judgment of the Investigator, would preclude scheduled study visits, completion of the study, or a safe administration of investigational product.
* Other protocol-specified exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 559 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2022-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Velazquez-Martin, MD, Study Director — Kodiak Sciences Inc
Locations (75):
- United States (59):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Northwest Arkansas Retina Associates, Springdale, Arkansas
  - California Retina Consultants, Bakersfield, California
  - Retina Vitreous Associates, Beverly Hills, California
  - Eye Medical Center of Fresno, Fresno, California
  - Retina Consultants of Orange County, Fullerton, California
  - UCSD Jacobs Retina Center, La Jolla, California
  - Retina Associates of Orange County, Laguna Hills, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Retina Consultants of San Diego, Poway, California
  - Retinal Consultants Medical Group Inc, Sacramento, California
  - Orange County Retina Medical Group, Santa Ana, California
  - California Retina Consultants, Santa Maria, California
  - Colorado Retina Associates PC, Lakewood, Colorado
  - Florida Eye Microsurgical Institute, Boynton Beach, Florida
  - Rand Eye Institute, Deerfield Beach, Florida
  - Retina Health Center, Fort Myers, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Retina Associates of Florida, Tampa, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates PA, Lenexa, Kansas
  - Vitreo Retinal Consultants and Surgeons, Wichita, Kansas
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Cumberland Valley Retina Consultants PC, Hagerstown, Maryland
  - New England Retina Consultants, Springfield, Massachusetts
  - Vitreo Retinal Associates PC, Worcester, Massachusetts
  - Foundation for Vision Research, Grand Rapids, Michigan
  - Associated Retinal Consultants PC, Royal Oak, Michigan
  - Vitreoretinal Surgery PA, Edina, Minnesota
  - Springfield Clinic LLP, Springfield, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - The Retina Center of New Jersey, Bloomfield, New Jersey
  - NJ Retina, Teaneck, New Jersey
  - Retina Associates of Cleveland, Beachwood, Ohio
  - Retina Associates of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cole Eye Institute, Cleveland, Ohio
  - Retina and Vitreous Center of Southern Oregon PC, Ashland, Oregon
  - Cascade Medical Research Institute, Eugene, Oregon
  - Retina Northwest, Portland, Oregon
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Palmetto Retina Center, Florence, South Carolina
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Southeastern Retina Associates PC, Knoxville, Tennessee
  - Tennessee Retina PC, Nashville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Austin Clinical Research, LLC, Austin, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Consultants of Texas (Katy), Katy, Texas
  - Texas Retina Associates, Plano, Texas
  - Austin Retina Associates (Round Rock), Round Rock, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Consultants of Texas (Woodlands), The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
- Axon Clinical, s.r.o., Prague, Czechia
- Germany (4):
  - Universitätsklinikum Bonn, Bonn
  - Uniklinik Köln, Cologne
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Leipzig, Leipzig
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga Eastern Clinical University Hospital Clinic Bikernieki, Riga
- Poland (3):
  - Oftalmika Sp. z o.o., Bydgoszcz
  - Gabinet Okulistyczny prof. E. Wylegala, Katowice
  - Retina Okulistyka Sp. z o.o. Sp. km., Warsaw
- Slovakia (4):
  - Univerzitna nemocnica Bratislava, Bratislava
  - Nemocnica Trebisov - SVET ZDRAVIA - PPDS, Trebišov
  - Fakultna nemocnica Trencin, Trenčín
  - Fakultna nemocnica s poliklinikou Zilina, Žilina
- Spain (2):
  - Institut de La Macula i La Retina, Barcelona
  - Hospital dos de Maig, Barcelona

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 72 medical centers between September 2019 and November 2020. The first participant was enrolled on 08 October 2019 and the last on 24 November 2020.
Pre-assignment Details: Of 785 participants screened, 559 were randomized to treatment. Two randomized subjects (one subject in KSI-301 arm and one subject in aflibercept arm) never received treatment, so do not have reason for not completing treatment.
Groups:
- KSI-301 5 mg Q12W-Q20W: Participants randomized to this arm received 5 milligrams (mg) KSI-301 intravitreal (IVT) injections once every 4 weeks (Q4W) to Week 8, followed by 5 mg KSI-301 IVT injections based on disease activity assessments and may vary from Q12W to Q20W until Week 52.
- Aflibercept 2 mg Q8W: Participants randomized to this arm received 2 milligrams (mg) aflibercept intravitreal (IVT) injections Q4W to Week 8, followed by 2 mg aflibercept IVT injections Q8W to Week 52.
Period: Overall Study
Arm/Group | KSI-301 5 mg Q12W-Q20W | Aflibercept 2 mg Q8W
Started | 277 (One participant did not receive any treatment.) | 280 (One participant did not receive any treatment.)
Completed (Completed is defined as participants who completed treatment through Year 1.) | 240 | 254
Not Completed | 37 | 26
Not completed — Adverse Event | 16 | 9
Not completed — Non-compliance with study drug | 0 | 3
Not completed — Withdrawal by Subject | 6 | 10
Not completed — Lost to Follow-up | 2 | 2
Not completed — Progressive disease | 11 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Patient moved out of state | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized subjects who received at least one active study treatment (KSI-301 or aflibercept)
Groups:
- Total: Total of all reporting groups
Arm/Group | KSI-301 5 mg Q12W-Q20W | Aflibercept 2 mg Q8W | Total
Number analyzed (Participants) | 277 | 280 | 557
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 23 | 41
  >=65 years | 259 | 257 | 516
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.6 (7.35) | 76.2 (8.27) | 76.4 (7.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 168 | 346
  Male | 99 | 112 | 211
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 9 | 26
  Not Hispanic or Latino | 260 | 271 | 531
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 271 | 272 | 543
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  North America | 229 | 235 | 464
  Europe | 48 | 45 | 93
BCVA in the Study Eye, Letters [Mean (Standard Deviation); unit: Letters] | 63.6 (12.23) | 63.6 (12.34) | 63.6 (12.27)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in BCVA in the Study Eye Averaged Over Weeks 48 and 52, Full Analysis Set Year 1
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity.
Time Frame: Year 1
Population: Full analysis set defined as all randomized subjects who received at least one treatment injection in Year 1. Subjects will be analyzed according to their randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: ETDRS Letters
Arm/Group | KSI-301 5 mg Q12W-Q20W | Aflibercept 2 mg Q8W
Number analyzed (Participants) | 277 | 280
ETDRS Letters | 1 (0.78) | 7 (0.77)
Statistical Analysis 1: Comparison: KSI-301 5 mg Q12W-Q20W vs Aflibercept 2 mg Q8W; Test type: Non-Inferiority — The maximum clinically acceptable true difference between KSI-301 and aflibercept participants to be considered non-inferior is 4 ETDRS letters, i.e. the non-inferiority margin (NI) is 4 letters; p > 0.9999, Mixed Models Analysis; MMRM model with treatment, visit, treatment by visit interaction, categories for baseline BCVA, BCVA-low luminance VA baseline, geographical location; Adjusted mean difference = -6.0, 95.03% CI 2-sided [-8 to -4], Standard Error of Mean 1.01

2. Secondary Outcome: Percentage of Subjects on KSI-301 Arm With a Once Every 12-Weeks, 16-Weeks or 20-Weeks Treatment Interval
Description: Percentage of subjects on KSI-301 arm achieving a Once Every 12-Weeks, 16-Weeks or 20-Weeks Treatment Interval based on individualized treatment response
Time Frame: Year 1
Population: Subjects with Available Data at the Planned Durability Assessment at Year 1
Measure: Count of Participants; unit: Participants
Groups:
- KSI-301 5 mg: Drug: KSI-301 5 mg. KSI-301 5 mg will be administered by intravitreal injection into the study eye at 12, 16, and 20 weeks intervals as specified in the study protocol.
  Drug: Sham Procedure. The sham is a procedure that mimics an intravitreal injection. It involves pressing the blunt end of an empty syringe (without a needle) against the anesthetized eye. It will be administered to participants in both treatments arms at applicable visits to maintain masking.
  KSI-301: Intravitreal Injection
  Sham Procedure: The sham is a procedure that mimics an intravitreal injection. It involves pressing the blunt end of an empty syringe (without a needle) against the anesthetized eye. It will be administered to participants in both treatments arms at applicable visits to maintain masking.
Arm/Group | KSI-301 5 mg
Number analyzed (Participants) | 234
Participants
  Number of participants on the KSI-301 Q12W | 71
  Number of participants on the KSI-301 Q16W | 24
  Number of participants on the KSI-301 Q20W | 139

3. Secondary Outcome: Percentage of Subjects Gaining ≥ 5, ≥10 and ≥15 Letters in BCVA From Baseline in the Study Eye, Full Analysis Set Year 1
Description: Categorical improvements in Best Corrected Visual Acuity (BCVA) of clinically relevant BCVA measurements corresponding to 1, 2 and 3 lines of the ETDRS vision testing chart
Time Frame: Year 1
Population: All randomized subjects who received at least one treatment injection in Year 1 with available data at Year 1 for analysis. Number of participants in each Row Title is not mutually exclusive as number of participants who gained >=15 ETDRS letters includes participants who gained >=10 ETDRS letters and participants who gained >=5 ETDRS letters.
Measure: Count of Participants; unit: Participants
Groups:
- Aflibercept 2 mg: Drug: Aflibercept 2 mg. Aflibercept 2 mg will be administered by intravitreal injection into the study eye once every 4 weeks for 3 consecutive months, followed by once every 8 weeks.
  Drug: Sham Procedure. The sham is a procedure that mimics an intravitreal injection. It involves pressing the blunt end of an empty syringe (without a needle) against the anesthetized eye. It will be administered to participants in both treatments arms at applicable visits to maintain masking.
  Aflibercept: Intravitreal Injection
  Sham Procedure: The sham is a procedure that mimics an intravitreal injection. It involves pressing the blunt end of an empty syringe (without a needle) against the anesthetized eye. It will be administered to participants in both treatments arms at applicable visits to maintain masking.
Arm/Group | KSI-301 5 mg | Aflibercept 2 mg
Number analyzed (Participants) | 238 | 254
Participants
  Gain >=5 ETDRS Letters at Year 1 | 103 | 148
  Gain >=10 ETDRS Letters at Year 1 | 66 | 87
  Gain >=15 ETDRS Letters at Year 1 | 31 | 46

4. Secondary Outcome: Percentage of Subjects Who Achieving BCVA Snellen Equivalent of 20/40 or Better in the Study Eye at Year 1
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. BCVA Snellen equivalent of 20/40 was defined as ≥69 ETDRS letters
Time Frame: Year 1
Population: All randomized subjects who received at least one treatment injection in Year 1 with available data at Year 1 for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 5 mg Q12W-Q20W | Aflibercept 2 mg Q8W
Number analyzed (Participants) | 238 | 254
Participants | 119 | 165

5. Secondary Outcome: Percentage of Subjects With BCVA Snellen Equivalent of 20/200 or Worse in the Study Eye at Year 1
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. BCVA Snellen equivalent of 20/200 or Worse was defined as BCVA ≤ 38 ETDRS Letters.
Time Frame: Year 1
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 5 mg Q12W-Q20W | Aflibercept 2 mg Q8W
Number analyzed (Participants) | 238 | 254
Participants | 13 | 8

6. Secondary Outcome: Mean Change in OCT Central Subfield Retinal Thickness (CST) From Day 1
Description: Central subfield thickness (CST) was defined as the distance between the internal limiting membrane (ILM) and the retinal pigment epithelium (RPE) as assessed by a central reading center.
Time Frame: Year 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | KSI-301 5 mg Q12W-Q20W | Aflibercept 2 mg Q8W
Number analyzed (Participants) | 277 | 280
Microns | -96.1 (123.39) | -134.1 (111.17)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) reported through Week 52 or Early Termination (ET) if occurred before Week 52.
Description: Safety results for the KSI-301 5mg arm are presented together as patients treated with Q12W dosing received 6 total doses in Year 1 and the patients treated with Q20W dosing received 5 total doses in Year 1. Therefore, presenting all treatment intervals together provides a more robust dataset to evaluate the safety profile of KSI-301.
Arm/Group | KSI-301 5 mg Q12W-Q20W | Aflibercept 2 mg Q8W
All-Cause Mortality (participants affected / at risk) | 4/277 | 8/280
Serious Adverse Events (participants affected / at risk) | 35/277 | 33/280
Other Adverse Events (participants affected / at risk) | 82/277 | 84/280
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KSI-301 5 mg Q12W-Q20W (N=277) | Aflibercept 2 mg Q8W (N=280)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Endophthalmitis - Study eye (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (4)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (3) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Retinal haemorrhage - Study eye (Eye disorders) | 2 (2) | 0 (0)
Neovascular age-related macular degeneration - Study eye (Eye disorders) | 1 (1) | 0 (0)
Rhegmatogenous retinal detachment - Study eye (Eye disorders) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ilium fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Perforated ulcer (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 3 (3)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Prostatic varices (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KSI-301 5 mg Q12W-Q20W (N=277) | Aflibercept 2 mg Q8W (N=280)
Neovascular age-related macular degeneration - Fellow eye (Eye disorders) | 19 (19) | 26 (26)
Retinal haemorrhage - Study eye (Eye disorders) | 17 (18) | 4 (5)
Cataract - Study eye (Eye disorders) | 15 (15) | 10 (10)
Conjunctival haemorrhage - Study eye (Eye disorders) | 13 (14) | 24 (30)
Urinary tract infection (Infections and infestations) | 15 (18) | 16 (18)
Hypertension (Vascular disorders) | 15 (15) | 16 (16)

LIMITATIONS AND CAVEATS:
This study was terminated early by the Sponsor because the study did not meet the primary endpoint. Thus, not all participants in this study completed the full duration of treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/66/NCT04049266/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT04049266/SAP_001.pdf